CLINICAL TRIAL: NCT06186765
Title: Prospective, Non-randomized, Multicenter Clinical Evaluation of the Recharge Free Axonics SNM System (Model 4101)
Brief Title: F15 Recharge Free Axonics SNM System Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Axonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105-0108
Record Dates: First submitted 2023-12-13; First posted 2024-01-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Urinary Urge Incontinence (UUI); Urinary Frequency (UF); Fecal Incontinence (FI)
MeSH Terms: conditions — Urinary Incontinence, Urge; Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm - product does not have Communauté Européenne (CE) Mark in Europe (Other): Observational
  Interventions: Device: Axonics SNM System (Model 4101)

INTERVENTIONS:
Device: Axonics SNM System (Model 4101) — Safety and performance/effectiveness assessment of the recharge free Axonics SNM System (Model 4101 in participants with overactive bladder (OAB) or fecal incontinence (FI).

SUMMARY:
Multicenter, prospective, non randomized, single arm evaluation of patients with overactive bladder (OAB) and/or fecal incontinence (FI) employing the Axonics recharge free SNM System.

DETAILED DESCRIPTION:
A clinical evaluation to comply with new European Medical Device Regulations (EU MDR) guidelines. Multicenter, prospective, non-randomized, single arm study for OAB and/or FI to assess the safety and performance of the Food and Drug Administration (FDA) approved Axonics recharge free sacral neuromodulation (SNM) System, INS Model 4101. The product is currently marketed under the name F15.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Primary indication of overactive bladder (OAB) (urinary urgency incontinence (UUI)/ urinary frequency (UF)) or fecal incontinence (FI) who are not candidates for, or who have failed conservative treatment
3. Willing and capable to provide written informed consent and agrees to comply with specified evaluations at clinical investigational sites and attend all follow-up assessments for up to 1 year.

Exclusion Criteria:

1. Any significant medical condition that is likely to interfere with procedures, device operation, or likely to confound evaluation of endpoints (exclusion of neurological conditions such as multiple sclerosis)
2. Any psychiatric or personality disorder that is likely to interfere with procedures at the discretion of the participating physician; this may include poor understanding or compliance with requirements
3. Previously underwent an external sacral neuromodulation (SNM) trial and was deemed a non-responder or was previously implanted with a sacral neuromodulation device and did not get therapeutic benefit (a non-responder)
4. History of allergic response to titanium, zirconia, polyurethane, epoxy, or silicone
5. A female who is breastfeeding
6. A female with a positive urine pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Performance/Effectiveness - Improvement in Quality of Life scoring (OAB) | 3 months
  International Consultation on Incontinence Questionnaire Overactive Bladder Quality of Life (ICIQ-OABqol): questions in each subscale are scored by a summed range of 0 to 100, with a higher score indicating better quality of life. Overall score ≥ 10 points from baseline to follow-up is indicative of a clinically meaningful improvement.
Performance/Effectiveness - Improvement in Fecal Incontinence Survey | 3 months
  Cleveland Clinic Florida - Fecal Incontinence Score (CCF-FIS): includes 5 items (solid, liquid, gas, wears pad and lifestyle alteration) and 5 frequencies (never = 0, rarely = 1, sometimes = 2, usually = 3, always = 4). Scores range from 0 for full continence to 20 for complete incontinence. A higher score is indicative of the severity of fecal incontinence.
Adverse event reporting (Safety) | 3 months
  Device-related, procedure-related and all serious adverse events

SECONDARY OUTCOMES:
Performance/Effectiveness - Improvement in Quality of Life scoring (OAB) | 1 year
  International Consultation on Incontinence Questionnaire Overactive Bladder Quality of Life (ICIQ-OABqol): questions in each subscale are scored by a summed range of 0 to 100, with a higher score indicating better quality of life. Overall score ≥ 10 points from baseline to follow-up is indicative of a clinically meaningful improvement.
Performance/Effectiveness - Improvement in Fecal Incontinence Survey | 1 year
  Cleveland Clinic Florida - Fecal Incontinence Score (CCF-FIS): includes 5 items (solid, liquid, gas, wears pad and lifestyle alteration) and 5 frequencies (never = 0, rarely = 1, sometimes = 2, usually = 3, always = 4). Scores range from 0 for full continence to 20 for complete incontinence. A higher score is indicative of the severity of fecal incontinence.
Performance/Effectiveness - Improvement in Quality of Life Survey (FI) | 3 months, 6 months, 1 year
  Fecal Incontinence Quality of Life (FIQoL): includes four different subscales: lifestyle, coping/behavior, depression/self-perception and embarrassment. Subscale scores range from 1 to 5, with 1 indicating lower functional status of qualify of life.
Adverse event reporting (Safety) | 1 year
  Device-related, procedure-related and all serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Bertil Blok, MD, PhD, Principal Investigator — Erasmus Medical Center; Gita Ghadimi, OD, Study Director — Boston Scientific Corporation
Locations (16):
- United States (11):
  - Hartford Healthcare, Waterford, Connecticut
  - Florida Gulf Clinical Research, Bradenton, Florida
  - East Coast Institute of Research, Jacksonville, Florida
  - Florida Bladder Institute, Naples, Florida
  - Atrium Health, Macon, Georgia
  - Minnesota Urology, Coon Rapids, Minnesota
  - Adult Pediatric Urology & Urogynecology, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York
  - The Oregon Clinic, Portland, Oregon
  - Southern Shores Urogynecology, Myrtle Beach, South Carolina
  - Houston Colon, Houston, Texas
- Erasmus Medical Center, Rotterdam, Netherlands
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Urological Institute, Bristol
  - University College London Hospital, London
  - Northern General Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No